CLINICAL TRIAL: NCT02816190
Title: PROne POsition and Volumetric CAPnography
Acronym: PROPOCAP
Status: Completed | Type: Observational
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Sebastien Jochmans, MD, ICU MD, Clinical Research Unit Director, Hopital of Melun
Other Study IDs: PROPOCAP
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Prone Position; Mechanical Ventilation; Volumetric Capnography
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: prone position

SUMMARY:
Beneficial effect of prone position in ARDS on mortality is not linked to increase in PF ratio. It is probably due to improvement in ventilation-perfusion ratio (V/Q). Volumetric capnography allows assessment of dead space and homogeneity of V/Q. All prone positionned patients will be included in the study with usual monitoring (i.e. respiratory system basic mechanics, volumetric capnography, blood gas samples). Epidemiologic and monitoring data will be collected during all prone position sessions.

ELIGIBILITY:
Inclusion Criteria:

* all prone positioned patients

Exclusion Criteria:

* age below 18 y, dependant patients, participation reject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All prone positionned patients
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
P3Slp | 24 hours
  Evolution of phase 3 slope of volumetric capnography in survivors vs non-survivors

CONTACTS AND LOCATIONS:
Overall Officials: sebastien jochmans, MD, Study Director — Clinical Research Unit, Melun Hospital
Locations (1):
- Melun Hospital ICU, Melun, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jochmans S, Mazerand S, Chelly J, Pourcine F, Sy O, Thieulot-Rolin N, Ellrodt O, Mercier Des Rochettes E, Michaud G, Serbource-Goguel J, Vinsonneau C, Vong LVP, Monchi M. Duration of prone position sessions: a prospective cohort study. Ann Intensive Care. 2020 May 24;10(1):66. doi: 10.1186/s13613-020-00683-7. PMID 32449068